CLINICAL TRIAL: NCT05449873
Title: No-touch Radiofrequency Ablation for Recurrent Hepatocellular Carcinoma After Locoregional Treatment Using Combined Energy Delivery Mode and Triple Cooled-Wet Electrodes
Brief Title: No-touch Radiofrequency Ablation for Recurrent Hepatocellular Carcinoma Using Triple Cooled-Wet Electrodes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: RF medical (Unknown)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2107-087-1235
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Recurrent Hepatocellular Cancer; Chronic Liver Disease and Cirrhosis
Keywords: No-touch radiofrequency ablation; Combined energy delivery mode; Triple cooled-wet electrodes
MeSH Terms: conditions — Liver Neoplasms; Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with recurrent hepatocellular carcinoma after locoregional treatment (Experimental): Patients with chronic liver disease have recurrent hepatocellular carcinoma which is diagnosed on contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI).
  Interventions: Procedure: Radiofrequency ablation using combined bipolar and monopolar energy deliver with Triple Cooled-Wet electrodes

INTERVENTIONS:
Procedure: Radiofrequency ablation using combined bipolar and monopolar energy deliver with Triple Cooled-Wet electrodes — Radiofrequency ablation will be performed by using triple cooled-wet electrodes. Two or three electrodes will be places around the tumor under ultrasonography (US)-computed tomography (CT)/magnetic resonance (MR) fusion tool guidance. The electrodes will be cooled with saline, and radiofrequency (RF, bipolar mode and switching monopolar mode) will be applied to two of three electrodes at the same time for about 6 to 30 minutes depending on the tumor size. The temperature will be maintained at 90-100 °C.

SUMMARY:
To evaluate local tumor progression rate at 12 months after no-touch percutaneous radiofrequency ablation using combined energy delivery mode and triple cooled electrodes

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh Class A or B
* chronic hepatitis B or chronic hepatitis C or liver cirrhosis
* presence of recurrent hepatocellular carcinoma (HCC) after locoregional treatment confirmed by pathology or imaging studies including contrast enhanced computed tomography (CT) or magnetic resonance imaging (MRI) according to Liver Imaging Reporting and Data System (LI-RADS) v2018
* single lesion less than or equal to 5 cm, or up to 3 lesions, each greater than less than or equal to 3 cm at the time of locoregional treatment

Exclusion Criteria:

* number of recurrent HCCs, equal or more than 3
* largest recurrent HCC size over 3 cm
* presence of vascular invasion by HCC
* platelet count less than 40,000 per mm3 or International Normalized Ratio (INR) prolongation over 50%
* presence of extrahepatic metastasis

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Local tumor progression rate | 12 months after radiofrequency ablation
  Evaluate local tumor progression by follow-up computed tomography (CT) or magnetic resonance imaging (MRI) with alpha-fetoprotein (AFP) level

SECONDARY OUTCOMES:
Disease-free survival | 12 moths after radiofrequency ablation
  Evaluate disease-free survival by available clinical information and follow-up computed tomography or magnetic resonance imaging with alpha-fetoprotein level
Technical success rate | 1 month after radiofrequency ablation
  Evaluate technical success defined as complete ablation of the index tumor with safety margin, equal or larger than 3 mm on 1 month follow-up CT.
Overall survival | 12 moths after radiofrequency ablation
  Evaluate overall survival by available clinical information and follow-up
Complication rate | 1, 3, 6, 9, 12 months after radiofrequency ablation.
  Evaluate the presence of major or minor radiofrequency ablation related complications on follow-up computed tomography or magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No